CLINICAL TRIAL: NCT07257783
Title: Effect of Buteyko Breathing Exercise Combined With Postural Stability Exercises on Maximal Oxygen Consumption in Young Adult Smokers
Acronym: BBE PSE VO2max
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yasmeen Alaa Abd El-Hamied Ahmeed (Other)
Responsible Party: Sponsor-Investigator, Yasmeen Alaa Abd El-Hamied Ahmeed, Teaching Assistant at Department of Physical Therapy for Internal Medicine & Geriatrics Faculty of Physical Therapy, Nahda University, Beni Suef, Egypt, October 6 University
Organization: October 6 University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: O6U.P.T.REC/024/003002; O6U.P.T.REC/024/003002 (Registry Identifier: october 6 university)
Record Dates: First submitted 2025-11-17; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Smoking ( Cigarette)
Keywords: Buteyko breathing exercise; Postural stability exercises; maximal oxygen consumption; young adult smokers
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: Treatment group and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): smokers didn't receive any intervention just measurement at the start of the study and at the end of the study
- study group (Experimental): Buteyko breathing exercise combined with postural stability exercises
  Interventions: Other: Buteyko breathing exercise combined with postural stability exercises

INTERVENTIONS:
Other: Buteyko breathing exercise combined with postural stability exercises — BBE: The therapist instructs the patient to sit comfortably, breathing naturally through the nose. They should hold their breath until the need to inhale arises, then exhale through the nasal passage. The patient maintains a straight back with feet shoulder-width apart, eyes closed, breathing calmly. After 20-30 seconds, they repeat the exercises for 3 minutes, followed by another pause and repetition. This is done for another 3 minutes, ending with a 2-minute rest before the next session. Duration: 15 minutes. PSE :Warming up phase: shoulder circles and twist torso during walking for 5 minutes. Training phase include 10-15 reps per set, 2-4 sets per exercise,30-60 seconds rest period between sets. Cooling down phase includes hold each stretch for 15-30 seconds, 2-4 reps per per side and rest for 15-30 seconds between reps. Bridging Side-lying leg raise Wall push-ups Lateral trunk flexion Chin tuck Stretch pectoralis major muscle,upper trapezius & SCM All these for 3/week for 6 weeks
  Arms: study group

SUMMARY:
Background: Smoking is one of the most significant risk factors for respiratory diseases, affecting both lung function and overall respiratory health. The harmful chemicals in tobacco smoke, contribute to airway inflammation, oxidative stress, and structural lung damage.

Purpose: The purpose of this study was to investigate effect of Buteyko breathing exercise combined with postural stability exercises on maximal oxygen consumption, pulmonary functions, oxygen saturation, functional capacity, and perceived exertion in young adult smokers. Subjects and procedures: Forty male smokers were recruit-ed from Nahda university. Their age ranged between 18-30 years. They were randomly assigned into 2 groups equal in number. Study Group: They participated in 6 weeks training with Buteyko breathing exercise combined with postural stability exercises (3 sessions per week) Control group: They weren't exposed to any intervention. Both groups were assessed by using pulse oximeter to measure oxy-gen saturation, Spirostilk to measure pulmonary functions, Borg scale to measure perceived exertion and six-minute walk test to measure functional capacity and maximal oxygen consumption.

ELIGIBILITY:
inclusion criteria

* Cigarette Smokers.
* Smoking period from 3 to 7 years
* They were medically stable.
* Age between 18 to 30 years.
* Male gender only was allowed to participate.
* They had the ability to perform exercises.
* Body mass index ranges from 21 to 25.

exclusion criteria

* Smokers diagnosed with any chronic disease or orthopedic problems.
* Mental disorders.
* Current intervention for cancer or active infection
* Obese their BMI above 26 and athlete people
* People who participated in any activity such as walking for long periods and swimming

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — In many populations, especially in developing countries, smoking is more common among men than women.This means:It's easier to recruit enough male participants & The sample better reflects the main smoking population To Avoid Hormonal and Biological Variability
Enrollment: 46 (Actual)
Dates: Start 2024-07-20 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
maximal oxygen consumption | From enrollment to the end of treatment at 6 weeks
  it is the highest rate at which the body can take in, transport, and utilize oxygen during intense exercise. It is considered a key indicator of cardiovascular fitness and endurance performance.
  Measured in: Milliliters of oxygen per kilogram of body weight per minute (ml/kg/min).
  it was calculated by estimated method from six minute walk test by this equation 12.701 + (0.06 × 6-minute walk distance m) - (0.732 × body mass indexkg/m2)

SECONDARY OUTCOMES:
oxygen saturation | From enrollment to the end of treatment at 6 weeks
  it refers to the percentage of hemoglobin molecules saturated with oxygen.Pulse oximetry is a simple, non-invasive, widely available medical tool that measures SpO2 through a device attached to a finger, a toe or an ear lobe.
forced viral capacity | From enrollment to the end of treatment at 6 weeks
  Spirometry was used to forced vital capacity (FVC)
perceived rate of exertion | From enrollment to the end of treatment at 6 weeks
  Measurement of PRE by Modified Borg scale It was used to rate how hard a person feels they are working from 0 to10 0 = No exertion at all & 10 = Maximal exertion
Functional capacity | From enrollment to the end of treatment at 6 weeks
  It was used to assess the cardiopulmonary fitness of the individuals. it is measured from 6-MWT
the ratio of forced expiratory volume in 1 Second to forced vital capacity | From enrollment to the end of treatment at 6 week
  Spirometry: was used to assess the ratio of forced expiratory volume in 1 Second (FEV₁) to forced vital capacity (FEV₁ /FVC)
forced expiratory volume in 1 Second | From enrollment to the end of treatment at 6 week
  Spirometry was used to assess forced expiratory volume in 1 Second (FEV₁)
Maximum voluntary ventilation | From enrollment to the end of treatment at 6 week
  Spirometry was used to assess maximum voluntary ventilation (MVV)

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy Nahda University, Banī Suwayf, Egypt